CLINICAL TRIAL: NCT00069134
Title: Glutathione Homeostasis and Oxidant Damage in Kwashiorkor
Brief Title: Study of Antioxidants and Oxidants in Malnourished Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Farook Jahoor, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLUTH - dk56689; R01DK056689 (NIH)
Record Dates: First submitted 2003-09-15; First posted 2003-09-17 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Protein-energy Malnutrition; Kwashiorkor; Marasmus
Keywords: glutathione kinetics; oxidant damage; anti-oxidant capacity; oxidative stress; cysteine kinetics; severe childhood malnutrition
MeSH Terms: conditions — Protein-Energy Malnutrition; Kwashiorkor | interventions — Amino Acids, Sulfur

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulfur Amino Acids (Experimental): 12 children with edematous severe malnutrition will be assigned to receive 0.65 mmol/kg/d of sulfur amino acids. Supplements will be added to the children's daily diets.
  Interventions: Dietary Supplement: sulfur amino acids
- Alanine (Placebo Comparator): 12 children with edematous severe malnutrition are assigned to receive 0.65 mmol/kg/d of alanine as placebo. Supplements will be added to the children's daily diets.
  Interventions: Dietary Supplement: sulfur amino acids

INTERVENTIONS:
Dietary Supplement: sulfur amino acids — Sixteen (16) children with edematous SCU will be randomly assigned to either a supplement of SAA or an isonitrogenous amount of alanine

SUMMARY:
It is believed that the organs of severely malnourished children malfunction because harmful compounds called oxidants injure the tissues in these organs. In a healthy person oxidants are made harmless because another compound called glutathione neutralizes them. Glutathione is made from three amino acids that we get from the protein we eat in our food. We found that malnourished children were not making enough glutathione because they lacked one of these amino acids called cysteine. In this study we determine why malnourished children do not have sufficient cysteine, and we will feed malnourished children a whey-based diet which is rich in cysteine during their treatment to determine whether they will make more glutathione. This in turn may make their organs recover faster. These findings will let us know whether malnourished children can recover faster if they are given more cysteine during the early phase of treatment.

ELIGIBILITY:
* Infants and toddlers, 6-18 months of age
* Suffering from severe protein-energy malnutrition, kwashiorkor and marasmic-kwashiorkor

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2003-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
small intestine, skin function and red blood cell gluathione synthesis | after intervention
  The effect of dietary supplementation with either a mixture of SAAs or alanine (controls) on:
  1. buccal tissue protein synthesis, small intestine structure, integrity and function (i.e. mixed mucosal and mucins protein synthesis rate, mucosal GSH synthesis and concentration, villous height and area and crypt depth, intestinal absorptive capacity and degree of mucosal leakiness, and synthesis of the starch digestive enzymes sucrase-isomaltase and maltase-glucoamylase, plus in vivo starch digestion and absorption) in groups of age- and gender-matched children with edematous SCU in the severely malnourished state.
  2. skin protein synthesis rate, rate of closure of skin lesions
  3. Red blood cell glutathione synthesis rate and cysteine production
immune capacity | after intervention
  synthesis rate of selected acute phase proteins

CONTACTS AND LOCATIONS:
Overall Officials: Farook Jahoor, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Tropical Metabolism Research Unit, University of the West Indies, Kingston, Saint Andrew Parish, Jamaica

REFERENCES:
- [Derived] Badaloo A, Hsu JW, Taylor-Bryan C, Green C, Reid M, Forrester T, Jahoor F. Dietary cysteine is used more efficiently by children with severe acute malnutrition with edema compared with those without edema. Am J Clin Nutr. 2012 Jan;95(1):84-90. doi: 10.3945/ajcn.111.024323. Epub 2011 Dec 14. PMID 22170355